CLINICAL TRIAL: NCT06623032
Title: Metabolic Effects of Medium-Chain Fatty Acids in Patients with Medium-Chain Acyl-CoA Dehydrogenase Deficiency and Healthy Individuals
Acronym: MEMCADD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Copenhagen Neuromuscular Center (Unknown); Center of Inherited Metabolic Diseases, Copenhagen University Hospital Rigshospitalet (Unknown); Section of Molecular Physiology, Department of Nutrition, Exercise and Sports, Faculty of Science, University of Copenhagen, Denmark (Unknown)
Responsible Party: Principal Investigator, Andreas Mæchel Fritzen, Associate Professor, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: H-24044278; NNF22OC0074110 (Other Grant/Funding Number: Novo Nordisk Foundation)
Record Dates: First submitted 2024-09-23; First posted 2024-10-02 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-10

CONDITIONS: Medium-chain Acyl-CoA Dehydrogenase Deficiency
Keywords: MCADD; Lipid metabolism; Ketone bodies; Medium-Chain Fatty Acid (MCFA); Long-Chain Fatty Acid (LCFA)
MeSH Terms: conditions — Medium chain acyl CoA dehydrogenase deficiency

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Healthy Participants (Experimental)
  Interventions: Other: Medium-Chain Fatty Acid (MCFA); Other: Long-Chain Fatty Acid (LCFA)
- MCADD Patients (Experimental)
  Interventions: Other: Medium-Chain Fatty Acid (MCFA); Other: Long-Chain Fatty Acid (LCFA)

INTERVENTIONS:
Other: Medium-Chain Fatty Acid (MCFA) — The participants will consume Medium-Chain Fatty Acid (MCFA) followed by Long-Chain Fatty Acid (LCFA)
Other: Long-Chain Fatty Acid (LCFA) — The participants will consume Long-Chain Fatty Acid (LCFA) followed by Medium-Chain Fatty Acid (MCFA).

SUMMARY:
The aim of this project is to investigate the physiological effects of intake of long-chain fatty acids (LCFA) and medium-chain fatty acids (MCFA) in patients with Medium-Chain Acyl-CoA Dehydrogenase Deficiency (MCADD) and healthy individuals

DETAILED DESCRIPTION:
Male and female MCADD patients and healthy individuals will be included in this study which is a randomized intervention study in a cross over design consisting of two separate test days.

The study involves two test days of four hours each, during which the participants ingests either medium-chain fatty acids (MCFA) or long-chain fatty acids (LCFA) in the form of triacylglycerol oils. The order of fatty acid oils ingested is determined by randomization.

ELIGIBILITY:
Inclusion Criteria MCADD patients:

* Male or female
* Age between 18-80 years old
* Diagnosed Medium-chain acyl-CoA dehydrogenase deficiency (MCADD

Inclusion Criteria Healthy Participants:

* Male or female
* Age between 18-80 years old

Exclusion Criteria both MCADD patients and healthy participants:

* Diabetes
* Kidney- or liver disease
* Use of beta blockers or diuretics
* Pregnant, lactating or planning to become pregnant within the study period
* Regular intake of substantial amounts of coconut oil, palm kernel oil or any other source abundant in MCFA
* Ongoing cancer treatment
* Metabolic or absorptive disorders, gastric bypass operation, or use of medication affecting metabolism or food absorption
* Inability, physically or mentally, to comply with the procedure required by the study protocol as evaluated by the primary investigator, study manager or clinical responsible

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-18 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Ketone Bodies | During both individual test days
  To measure the effect of Medium-Chain Fatty Acid (MCFA) and Long-Chain Fatty Acid (LCFA) on circulating ketone body concentrations.

SECONDARY OUTCOMES:
Resting metabolic rate | During both individual test days
  To measure the effect of Medium-Chain Fatty Acid (MCFA) and Long-Chain Fatty Acid (LCFA) on resting metabolic rate.
Respiratory exchange ratio | During both individual test days
  To measure the effect of Medium-Chain Fatty Acid (MCFA) and Long-Chain Fatty Acid (LCFA) on respiratory exchange ratio.
Vasodilator Function | During both individual test days
  To measure the effect of Medium-Chain Fatty Acid (MCFA) and Long-Chain Fatty Acid (LCFA) on vasodilator function.
Fatty Acid Composition | During both individual test days
  To measure the effect of Medium-Chain Fatty Acid (MCFA) and Long-Chain Fatty Acid (LCFA) on fatty acid composition.
Metabolites | During both individual test days
  To measure the effect of Medium-Chain Fatty Acid (MCFA) and Long-Chain Fatty Acid (LCFA) on circulating ketone body concentrations.
Hepatokines | During both individual test days
  To measure the effect of Medium-Chain Fatty Acid (MCFA) and Long-Chain Fatty Acid (LCFA) on circulating hepatokine concentrations.
Beta cell function | During both individual test days
  To measure the effect of Medium-Chain Fatty Acid (MCFA) and Long-Chain Fatty Acid (LCFA) on Beta cell function.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas M Fritzen, Associate Professor, Principal Investigator — University of Copenhagen
Locations (1):
- University of Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No